CLINICAL TRIAL: NCT01271647
Title: Randomized Controlled Trial of Classic Yin and Yang Tonic Formula in Osteopenia
Brief Title: Classic Yin and Yang Tonic Formula for Osteopenia
Acronym: CYYTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: yongjun wang, Shanghai UTCM
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LHCTOP2011
Record Dates: First submitted 2011-01-03; First posted 2011-01-07 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-01

CONDITIONS: Osteopenia
Keywords: osteopenia,chinese herb
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chinese herb (Experimental)
  Interventions: Drug: Yin and Yang tonic granules
- placebo (Experimental)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Yin and Yang tonic granules — Yin and Yang tonic granules,18g per time,two times per day,six months
  Other Names: Zuo and You gui Granules
  Arms: chinese herb
Drug: placebo — granules,18g per time,two times per day,six months
  Other Names: Zuo and You gui Granules
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the classic yin and yang tonic formula for osteopenia and to research the mechanism of efficacy.

DETAILED DESCRIPTION:
Osteoporosis is a growing problem worldwide, with the greatest burden resulting from fractures. Nevertheless, the majority of fractures in adults occur in those with "osteopenia" (bone mineral density (BMD) only moderately lower than young normal individuals) Since life long drug therapy is an expensive option with uncertain consequences and side effect, natural herbal therapy offers an attractive alternative. The classic Yin and Yang Tonic Formula (eg.Zuogui Pill, Yougui Pill) have been used for osteoporosis or osteopenia in traditional Chinese medicine(TCM) for a long time. For this reason, Chinese guidelines for the treatment of osteopenia include natural herbal therapy, however, there is currently no randomize placebo controlled trial to verify the efficacy for treating low BMD. This trial is randomized, double blind, placebo controlled design. Results of this study will provide evidence regarding the value of the classic Yin and Yang tonic formula as an intervention for increase BMD and decreasing fracture risk in osteopenia. Furthermore, the mechanisms of action can be identified by this study.

ELIGIBILITY:
Inclusion Criteria:

* BMD T-scores of the hip (femoral neck or trochanter)and/or spine between -1.0 and -2.5;
* pattern differentiation is kidney deficiency in TCM.
* informed consent.

Exclusion Criteria:

* Osteoporotic (T-score< -2.5) at any site or a fracture in the past 2 years not caused by motor vehicle accident;
* prior or current use of medication that increase risks of fracture (e.g. steroids, anti-convulsants, anticoagulants,lithium);
* prior or current use of medications that modify bone metabolism (e.g. bisphosphonates, selective estrogen receptor modulators such as Raloxifene);
* use of calcium supplements above levels suggested within the recommendations of standard care (i.e., above 1200-1500 mg);
* current or prior year use of estrogen or calcitonin;
* Malignancies other than skin cancer;
* conditions that cause secondary osteoporosis (e.g. Cushing's syndrome, Marfan's syndrome);
* lactation and gestational period;
* physical or mental disabilities that will preclude informed consent or active study participation;
* supersensitivity body constitution.
* osteoporotic fracture of having operating indication.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | 6 months

SECONDARY OUTCOMES:
pain visual analogue scales,ECOS-16 questionnaire,bone metabolism,NEI. | 6 months
  pain visual analogue scales:6month ECOS-16 questionnaire:6month bone metabolism,NEI:6month

CONTACTS AND LOCATIONS:
Overall Officials: feng yang, doctor, Study Director — Shanghai UTCM
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang F, Tang DZ, Cui XJ, Holz JD, Bian Q, Shi Q, Wang YJ. Classic yin and yang tonic formula for osteopenia: study protocol for a randomized controlled trial. Trials. 2011 Aug 2;12:187. doi: 10.1186/1745-6215-12-187. PMID 21806837